CLINICAL TRIAL: NCT03849105
Title: A Multi-centre, Open-label, Single-arm, Dose-finding Phase I/II Study to Evaluate Safety, Tolerability, Dosing Schedule, and Preliminary Efficacy of Carrier-added 4-L-[131I]Iodo-phenylalanine (131I-IPA), Administered as Single or Repetitive Injections in Patients With Recurrent Glioblastoma Multiforme (GBM), Concomitantly to 2nd Line External Radiation Therapy (XRT) - IPAX- 1
Brief Title: 131I-IPA and Concurrent XRT in Recurrent GBM
Acronym: IPAX-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131I-IPA-TLX-101-001
Record Dates: First submitted 2019-01-29; First posted 2019-02-21 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2021-11

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma multiforme (GBM),; External Radiotherapy; 131I-IPA
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: multi-centre, open-label, dose-finding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single administration of 131I-IPA (1f group) (Experimental): Study participants with GBM receive a single administration of 4-L-[131I]iodo-phenylalanine (131I-IPA), followed by 18 cycles of external radiotherapy, each cycle being of 2 Gy.
  Interventions: Radiation: 4-L-[131I]iodo-phenylalanine (131I-IPA)
- Three administrations of 131I-IPA (3f-parallel group) (Experimental): Study participants will be administered in 2GBq in 3 fractions corresponding to ⅓ full dose activity (0.67 GBq for the 2.0 GBq dose level). The 1st fraction of 131I-IPA will be administered as above, 1- 3 days prior to 1st XRT. The 2nd and 3rd 131I-IPA fractions will be administered after 5-9 XRT fractions (subject to investigator's discretion and day of IMP administration) following the previous 131I-IPA fraction. The remainder of XRT fractions will be given following the 3rd 131I-IPA fraction.
  Interventions: Radiation: 4-L-[131I]iodo-phenylalanine (131I-IPA)
- Three administrations of 131I-IPA (3f-sequential group) (Experimental): Study participants will be administered in 2GBq in 3 fractions corresponding to ⅓ full dose activity (0.67 GBq for the 2.0 GBq dose level). The 1st fraction of 131I-IPA will be administered as above 1- 3 days prior to 1st XRT. The 2nd 131I-IPA fraction will be administered after all 18 XRT fractions have been completed, and the 3rd 131I-IPA fraction will be administered 1 week after the 2nd 131I-IPA fraction.
  Interventions: Radiation: 4-L-[131I]iodo-phenylalanine (131I-IPA)
- Dose escalation of fractionated dosing (Experimental): Dose escalation will be made in steps of 2.0 GBq, i.e. 4.0 (3*1.33 GBq), 6.0 GBq (3*2.0 GBq), up to 8.0 GBq (3*2.67 GBq) until the maximum tolerated dose (MTD) is reached, using cohorts of N=3 patients.
  Interventions: Radiation: 4-L-[131I]iodo-phenylalanine (131I-IPA)

INTERVENTIONS:
Radiation: 4-L-[131I]iodo-phenylalanine (131I-IPA) — Study participants will receive by intravenous infusion an escalating activity of 4-L-[131I]iodo-phenylalanine (131I-IPA).
  Additional therapy is received in the form of externally administered radiotherapy
  Other Names: external radiotherapy

SUMMARY:
A multi-centre, open-label, single-arm, dose-finding phase I/II study to evaluate safety, tolerability, dosing schedule, and preliminary efficacy of carrier-added 4-L-[131I]iodo-phenylalanine (131I-IPA), administered as single or repetitive injections in patients with recurrent glioblastoma multiforme (GBM), concomitantly to 2nd line external radiation therapy (XRT) - IPAX-1

DETAILED DESCRIPTION:
The IPAX-1 study is an open-label, single-arm, randomised, parallel-group, multi-centre dose-finding study to evaluate ascending radioactive dose levels of 131I-IPA, intravenously administered using different dose schedules (fractionations), concomitantly to 2nd line XRT (36 Gy, administered in 18 fractions of 2 Gy). Gross tumour volume will be determined using contrast-enhanced MRI and amino acid-based PET imaging (18F-FET or 11C-methionine).

Patients will be included if they meet all of the following criteria:

1. Previously confirmed histological diagnosis of GBM, with current clinical or imaging evidence for first recurrence according to modified RANO criteria (2017). History of GBM standard therapy (debulking surgery, followed by radio-chemotherapy (50-60 Gy in 2 Gy fractions, temozolomide)
2. Interval since end of 1st line XRT ≥6 months
3. Amino acid-based molecular imaging (preferably 18F-FET- PETor 11C-methionine, as institutionally established) indicating pathologically increased amino acid uptake inside or in the vicinity of the tumour, clearly discernible from background activity.
4. Current indication for repeat radiation therapy as discussed at the multidisciplinary neuro-oncological tumour board meeting, planned as standard fractionated dose schedule (18*2 Gy)
5. Gross tumour volume (GTV) of up to 4.8 cm diameter, clinical target volume (CTV) 0.5 cm margin and planning target volume (PTV) less than or equal to 0.5 cm margin
6. Male or female ≥18 years of age.
7. Karnofsky performance status (KPS) ≥70. Life expectancy of at least 16 weeks.
8. Haematological, liver and renal function test results as follows:

   * WBC: >3*109/L
   * Haemoglobin >80 g/L
   * PLT >100*109/L
   * ALT, ALP, AST: ≤5 times upper international limit of normal (UILN)
   * Bilirubin ≤3 times UILN
   * Serum creatinine: within normal limits or <120 μmol/L for patients aged 60 years or older
   * Urine protein dipstick: no protein
9. Female patients surgically sterile or postmenopausal for at least 2 years. Participants of generative potential agreeing to use effective contraception during the period of therapy and 6 months after the end of study.
10. Written informed consent

A patient will be excluded from participation in the trial if one or more of the following criteria are met:

1. Primary XRT dose greater than 60 Gy
2. Doses to organs at risk defined by Yasar and Tugrul (2005) exceeded or reached by prior radiation therapy; e.g. cumulative total dose on the optical chiasm greater than 54 Gy for 2 Gy/fraction
3. Multifocal distant recurrence, defined as tumour lesion outside the primary XRT field, as evidenced by amino acid-based PET imaging
4. Prior treatment with brachytherapy
5. Prior treatment with bevacizumab
6. History or evidence of delayed-type hypersensitivity (DTH)-dependent chronic infection (e.g. tuberculosis, systemic fungal or parasitic infection), potentially exacerbating under systemic corticoid therapy
7. Localisation of tumour related to brain stem or axis, unless sufficient reserve capacity (e.g. remnant resection cavity, marked atrophy) to accommodate possible post- procedural tissue reactions, or pre-therapeutic consent for emergency trepanation
8. Haemostaseologic conditions, precluding catheterisation or invasive procedures
9. Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product
10. Known impairment of liver or kidney function or known liver or kidney disease, such as hepatitis, cirrhosis, renal failure
11. Known human immunodeficiency virus (HIV) positive serology or chronically active hepatitis B or C
12. Ongoing toxicity > grade 2 NCI-CTC (version 4.03) from previous standard or investigational therapies
13. Administration of another investigational medicinal product within 90 days prior to screening
14. Expected non-compliance with longer-term admission at isolated nuclear medicine ward
15. In pre-menopausal women: Pregnant as evidenced by a positive pregnancy test, or breast-feeding
16. Patients with known phenylketonuria

Study Design:

At the first dose level of 2 GBq, 131I-IPA will be administered in one of three different dosing regimens:

* Single dose regimen (1f group): Full 131I-IPA activity (2.0 GBq at the 2 GBq dose level) will be administered 1- 3 days prior to 1st XRT as a single injection.
* Fractionated dose regimen (3f - parallel group): 131I-IPA activity will be administered in 3 fractions corresponding to ⅓ full dose activity (0.67 GBq for the 2.0 GBq dose level). The 1st fraction of 131I-IPA will be administered as above, 1- 3 days prior to

  1st XRT. The 2nd and 3rd 131I-IPA fractions will be administered after 5-9 XRT fractions (subject to investigator's discretion and day of IMP administration) following the previous 131I-IPA fraction. The remainder of XRT fractions will be given following the 3rd 131I-IPA fraction.
* Fractionated dose regimen (3f - sequential group): 131I-IPA activity will be administered in 3 fractions corresponding to ⅓ full dose activity (0.67 GBq for the 2.0 GBq dose level). The 1st fraction of 131I-IPA will be administered as above 1- 3 days prior to 1st XRT. The 2nd 131I-IPA fraction will be administered after all 18 XRT fractions have been completed, and the 3rd 131I-IPA fraction will be administered 1 week after the 2nd 131I-IPA fraction. The 2nd and 3rd 131I-IPA injections should be given on the same day of the week, and some hours after administration of the respective XRT dose of that day. The day of IMP administration is subject to change at investigator's discretion. The three different treatment groups at the first (2.0 GBq) dose level (131I-IPA single dose 1f and 131I-IPA fractionated dose either 3f parallel or 3f sequential) will be recruited in parallel, as appropriate. Patients will be allocated to one of the three IPA dosing regimens. N=3 patients will be enrolled for each of the three treatment schedules. A 10th patient can be added to any of the three groups, in order to corroborate evidence for possible differences in safety and efficacy.

Patients at the entry dose level of 2 GBq will undergo 131I-IPA brain SPECT for tumour dosimetry (performed in all patients), whole body planar imaging for determination of biodistribution and whole body safety dosimetry. In addition, these patients will be comparatively assessed for possible differences in safety and/or efficacy among the different dosing regimens.

Dose escalation beyond 2 GBq will be made using the fractionated dosing regimen only, unless the outcome of the 2 GBq dose level suggests otherwise. The best treatment schedule (3f parallel or 3f sequential, see above) for higher doses shall be selected after completion of the 2 GBq dose level.

Dose escalation will be made in steps of 2.0 GBq, i.e. 4.0 (3*1.33 GBq), 6.0 GBq (3*2.0 GBq), up to 8.0 GBq (3*2.67 GBq) until the maximum tolerated dose (MTD) is reached, using cohorts of N=3 patients.

If MTD has not been reached at 8.0 GBq, dose escalation may further proceed, increasing the dose fractions to a total dose 131I- IPA greater than 8 GBq using cohorts of N=3 as follows: 10 GBq, 3f (i.e. 3*3.33 GBq); 12 GBq, 3f (i.e. 3*4 GBq), etc., until MTD is reached or until a satisfactory anti-neoplastic efficacy is observed.

For assessment of possible anti-neoplastic effects during dose escalation, only amino acid-based molecular imaging (preferably 18F-FET-PET) will be used, which allows assessment of treatment-induced changes based on a single post-therapeutic imaging study.

MTD is defined as the dose level, inducing dose limiting toxicity (DLT), in not more than 1/6 of the subjects receiving such dose. MTD will be determined on day 45 from the first IPA injection. DLT is defined as grade 4 neurotoxicity or any other grade 4 toxicity according to NCI-CTC (version 4.03). If DLT is observed in 1 subject of a cohort, 3 additional patients will be treated at the same dose level, under which such toxicity occurred. If one or more of these patients (i.e. 2/4, 2/5 or 2/6) experience grade 4 toxicity, MTD will have been exceeded for the respective dose level. In such a case, 3 additional patients will be treated at the preceding dose level. Therapy-induced early necrosis, (also termed pseudo-progression, which has been associated with improved survival will not be classified as DLT if asymptomatic, or if symptomatic and at least partially reversible within three months with or without therapy. Disease progression/PsPD will be diagnosed according to the current RANO criteria (2017).

The highest dose under which no more than 1/6 of the patients experience DLT will be declared the MTD level. Safety, tolerability and evidence of anti-tumour effects will be compared between all dose levels, in order to identify a most suitable dose level (MSDL) for the phase II part. The MSDL will not necessarily be identical to the MTD, but might be selected by jointly considering efficacy, safety and radiation protection aspects. The identification of the MSDL will be made by a Drug Data Safety Monitoring Board (DSMB), based on an integrated review of efficacy and safety from the first part. Based on a comprehensive analysis of the first part results, the DSMB will make a conclusion regarding safety and efficacy, and recommend to the sponsor a dosing strategy and dose level (MSDL) for the phase II part, if merited. Prior to initiating phase II, the sponsor commits to submit a substantial amendment, containing a summary of the phase I results to the Austrian BASG, other competent authorities, and the responsible Ethics Committee, as appropriate.

Upon establishment of the MSDL, 12-22 further patients will be treated at the MSDL (Phase II). If unequivocal evidence of efficacy is observed, another 10 patients shall be included in the phase II part. It is planned to include approximately 34 (22+12) patients with recurrent GBM with the option to extend phase II study by another 10 patients if the results are encouraging (22+22 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Previously confirmed histological diagnosis of GBM, with current clinical or imaging evidence for first recurrence according to modified RANO criteria (2017). History of GBM standard therapy (debulking surgery, followed by radio-chemotherapy (50-60 Gy in 2 Gy fractions, temozolomide)
2. Interval since end of 1st line XRT ≥6 months
3. Amino acid-based molecular imaging (preferably 18F-FET-PETor 11C-methionine, as institutionally established) indicating pathologically increased amino acid uptake inside or in the vicinity of the tumour, clearly discernible from background activity.
4. Current indication for repeat radiation therapy as discussed at the multidisciplinary neuro-oncological tumour board meeting, planned as standard fractionated dose schedule (18*2 Gy)
5. Male or female ≥18 years of age.
6. Karnofsky performance status ≥70. Life expectancy of at least 16 weeks.
7. Haematological, liver and renal function test results as follows:

   * WBC: >3*109/L
   * Haemoglobin >80 g/L
   * PLT >100*109/L
   * ALT, ALP, AST: ≤5 times upper international limit of normal (UILN)
   * Bilirubin ≤3 times UILN
   * Serum creatinine: within normal limits or <120 μmol/L for patients aged 60 years or older
   * Urine protein dipstick: no protein
8. Female patients surgically sterile or postmenopausal for at least 2 years. Participants of generative potential agreeing to use effective contraception during the period of therapy and 6 months after the end of study.
9. Written informed consent

Exclusion Criteria:

1. Primary XRT dose < 60 Gy
2. Doses to organs at risk defined by Yasar and Tugrul (2005) exceeded or reached by prior radiation therapy; e.g. cumulative total dose on the optical chiasm >54 Gy for 2 Gy/fraction, alphas/beta=2
3. Multifocal distant recurrence, defined as tumour lesion outside the primary XRT field, as evidenced by amino acid-based PET imaging
4. Prior treatment with brachytherapy
5. Prior treatment with bevacizumab
6. Baseline steroid requirement , exceeding physiologic replacement doses ( <1.5 mg dexamethasone or equivalent per day)
7. History or evidence of delayed-type hypersensitivity (DTH)-dependent chronic infection (e.g. tuberculosis, systemic fungal or parasitic infection), potentially exacerbating under systemic corticoid therapy
8. Localisation of tumour related to brain stem or axis, unless sufficient reserve capacity (e.g. remnant resection cavity, marked atrophy) to accommodate possible post-procedural tissue reactions, or pre-therapeutic consent for emergency trepanation
9. Haemostaseologic conditions, precluding catheterisation or invasive procedures
10. Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product
11. Known impairment of liver or kidney function or known liver or kidney disease, such as hepatitis, cirrhosis, renal failure
12. Known human immunodeficiency virus (HIV) positive serology or chronically active hepatitis B or C
13. Ongoing toxicity > grade 2 NCI-CTC (version 4.03) from previous standard or investigational therapies
14. Administration of another investigational medicinal product within 90 days prior to screening
15. Expected non-compliance with longer-term admission at isolated nuclear medicine ward
16. In pre-menopausal women: Pregnant as evidenced by a positive pregnancy test, or breast-feeding
17. Patients with known phenylketonuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameter Adverse Events | From first administration of 131I-IPA until 12 months after first administration
  Treatment-related adverse events according to NCI-CTCAE v 4.03 criteria will be captured and evaluated for each patient
Safety parameter heart rate | From first administration of 131I-IPA until 12 months after first administration
  Frequency of occurrence and severity of abnormal findings as measured by beats per minute
Safety parameter blood pressure | From first administration of 131I-IPA until 12 months after first administration
  Frequency of occurrence and severity of abnormal findings as measured by mmHg
Safety parameter Liver function test | From first administration of 131I-IPA until 12 months after first administration
  This outcome will be measured on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria. Results will be assessed by number of participants with abnormal laboratory values.
Safety parameter Renal function test | From first administration of 131I-IPA until 12 months after first administration
  This outcome will be measured on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria. Results will be assessed by number of participants with abnormal laboratory values.
Safety parameter Full Blood Count | From first administration of 131I-IPA until 12 months after first administration
  This outcome will be measured on all patients with treatment-related adverse events based on criteria as determined by the NCI CTCAE v 5.0 criteria. Results will be assessed by number of participants with abnormal laboratory values.

SECONDARY OUTCOMES:
To evaluate the maximum tolerated dose (MTD) of 131I -IPA administered concomitantly to 2nd line XRT in recurrent GBM 2 | Evaluation of patient up to 30 days after completion of study therapy
  MTD will be calculated in cohorts of 3 patients that are evaluated for treatment-related adverse events according to NCI-CTCAE v 4.03. Dose will be escalated until such time that treatment-related grade 3 adverse events occur.
To evaluate the efficacy of a fractionated administration of 131I-IPA | Up to 6 months after completion of study therapy
  This outcome will be evaluated by comparing morphological outcomes to treatment, as assessed by imaging, between two treatment groups. The first treatment group having the dose administered in a single administration, whilst the second group will have the dose administered in three administrations
Dosimetry | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  To evaluate the radiation absorbed dose to tumour from 131I-IPA
Dosimetry | Up to 30 days after completion of study therapy
  To confirm biodistribution and absorbed doses to whole body and organs from 131I-IPA
To explore the antineoplastic effect of 131I-IPA + XRT combination therapy | Commencing just prior to first administration of 131I-IPA until 12 months from time of first therapeutic administration
  This outcome will be determined in all patients by the use of sequential CT imaging in order to determine response of the lesion to the therapy according to RANO criteria.
To explore the occurrence and frequency of pseudo-progression (PP) in response to 131I-IPA + XRT combination therapy | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  This outcome will be determined in all patients by the use of sequential CT imaging in order to determine the presence of pseudo progression as defined by the RANO criteria response to 131I-IPA + XRT combination therapy
To explore the cognitive function of participants | Test will be adminsterd at baseline, 45 days post dose of 131I-IPA, Month 3 and Month 6
  This outcome will be determined in all patients through the use of the Trail Making Test
To explore the cognitive function of participants | Test will be adminsterd at baseline, 45 days post dose of 131I-IPA, Month 3 and Month 6
  This outcome will be determined in all patients through the use of the HVLT-R
To explore the cognitive function of participants | Test will be adminsterd at baseline, 45 days post dose of 131I-IPA, Month 3 and Month 6
  This outcome will be determined in all patients through the use of the MAE COWA test

CONTACTS AND LOCATIONS:
Overall Officials: Josef Pichler, MD, Principal Investigator — Kepler University Clinic, Linz, Austria; Tatjana Traub-Weidinger, Principal Investigator — Medical University of Vienna
Locations (5):
- Lake Macquarie Private Hospital, Gateshead, New South Wales, Australia
- Austria (2):
  - Kepler University Clinic, Linz
  - Medical University of Vienna, Vienna
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam
  - UMC Utrecht Cancer Center, Utrecht